CLINICAL TRIAL: NCT02582762
Title: Pilot Study of Efficacy of Nail Gel Containing Artemisia Abrotanum Extract and Glycerin in Finger Nail Surface Abnormality
Brief Title: Pilot Study of Efficacy of Nail Gel in Finger Nail Surface Abnormality
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 658/2557(EC1)
Record Dates: First submitted 2015-10-18; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Nail Abnormalities
Keywords: Nail gel; Nail surface abnormality; Efficacy
MeSH Terms: conditions — Nails, Malformed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nail gel (Experimental): apply nail gel twice daily
  Interventions: Drug: Nail gel

INTERVENTIONS:
Drug: Nail gel — apply nail gel on affected nails twice daily for 2 months
  Other Names: Locycare

SUMMARY:
Nail surface abnormalities is any conditions that affect the nail matrix or nail bed which cause nail plates grow defectively. Common nail surface abnormalities are pitting nails, longitudinal ridging, and transverse ridging/Beau's line. Aging nails usually have nail surface abnormalities as well.

Nail gels are artificial nails used widely for aesthetic purposes. Although, their cosmetic use is increasing with day by day, their usefulness in conditions such as nail biting, brittle nails, and ingrown toe nails has been reported. Moreover, a previous study reported the benefits of nail gels in terms of improving nail surface abnormalities like pitting nails, trachyonychia, and onychoschizia.

This study was conducted to evaluate the efficacy of nail gel containing Glycerin which has humectant effect and Artemisia Abrotanum extract which has anti-fungal/bacterial activities in finger nail surface abnormalities.

DETAILED DESCRIPTION:
Evaluation of nail surface abnormality can be done by using Visiometer® (bioengineering measurement) and dermoscope. Both techniques are non-invasive.

Artemisia Abrotanum extract has been used as ingredient in cosmetic products and its safety has been declared. Undesirable events from external using products containing this substance have never been reported yet. Nail gel product in this study has been approved as a cosmetic product by Food and Drug Administration of Thailand (Thai FDA).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or above
2. Being diagnosed nail surface abnormalities stably more than 3 months

Exclusion Criteria:

1. Having severe or uncontrolled concomitant diseases
2. Having nail infection
3. History of manicure within the last 1 month
4. Use of Biotin or other nail modifying drugs within the previous 3 months
5. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Improvement overall nail surface abnormalities | 2 weeks and 8 weeks
  Number of nails of each participant with change/improvement nail surface using clinical assessment

SECONDARY OUTCOMES:
Improvement roughness of nail surface abnormalities | 2 weeks, and 8 weeks
  Number of nails of each participant with change/improvement nail surface using bioengineering measurement
Increase nail hydration | 2 weeks, and 8 weeks
  Number of nails of each participant with the increase of nail hydration using bioengineering measurement
Patients's satisfaction | 2 weeks and 8 weeks
  good patients's satisfaction outcome by self-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sumanas Bunyaratavej, MD, Principal Investigator — Siriraj Hospital, Mahiidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Bangkoknoi, Thailand